CLINICAL TRIAL: NCT00213317
Title: Could Lumbo-sacral Magnetic Stimulation Modify Recto-colonic Motility?
Brief Title: Effect of Lumbo-sacral Magnetic Stimulation on Colonic Motility
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2003/041/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Functional Colonic Disease; Fecal Incontinence
Keywords: sacral magnetic stimulation; fecal incontinence; constipation
MeSH Terms: conditions — Colonic Diseases, Functional; Fecal Incontinence; Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: lombo-sacral magnetic stimulation — repetitive lombo-sacral nerve magnetic stimulation active and placebo performed during colonic recordings after bisacodyl instillation

SUMMARY:
The purpose of this study is to evaluate the effect of sacral nerve magnetic stimulation on the colonic motility in healthy subjects, in incontinent and constipated patients.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers

Exclusion Criteria:

pregnant women metallic material implanted organic digestive disease neuro-surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers without anorectal or neurological disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie LEROI, PHD, Principal Investigator — University Hospital, Rouen